CLINICAL TRIAL: NCT06596330
Title: Integration of a Trained Language Model to Improve Glycemic Control Through Increased Physical Activity: a Fully Digital My Heart Counts Smartphone App Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel Seung Kim, Fellow in Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 76338
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Type2diabetes
MeSH Terms: interventions — Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LLM-generated coaching prompt (Experimental)
  Interventions: Behavioral: Validation of language model prompts in increasing short-term physical activity; Behavioral: Assessment of long-term changes to physical activity and glycemic control
- 10,000 Step Reminder (Active Comparator)
  Interventions: Behavioral: Validation of language model prompts in increasing short-term physical activity; Behavioral: Assessment of long-term changes to physical activity and glycemic control

INTERVENTIONS:
Behavioral: Validation of language model prompts in increasing short-term physical activity — Aim 1: In preliminary data, the investigators have pre-trained an open-source language model, LLAMA, with expert-created coaching prompts based on the stages of change model for physical activity. Seven different prompts (for each day of an intervention "week") will be generated, accounting for race/ethnicity, age, gender, and stage of change, to improve personalization. Using the existing MHC app, the investigators will perform a randomized crossover trial on mean daily steps across each intervention. The investigators will compare the interventions of a daily reminder to reach 10,000 steps (a neutral control) and AI-personalized interventions based on an individual's stage of change.
Behavioral: Assessment of long-term changes to physical activity and glycemic control — Aim 2: Using social accountability and the trained language model generating personalized coaching interventions, the investigators will conduct a long-term follow-up randomized, unblinded trial. Over a 24-week intervention period, participants will receive either a generic daily reminder to reach 10,000 steps or an AI-generated coaching prompt, with the AI group also being able to "chat" with the language model to ask for advice on maintaining their physical activity. The outcomes of this long-term trial will be change in: 1) daily steps over the intervention period, 2) weight (via HealthKit link to MHC), and 3) HbA1c (as derived from EMR records linked to the HIPAA-compliant MHC app).

SUMMARY:
Type 2 diabetes (T2D) is one of the most common and fastest growing diseases, affecting 1 in 8 adults (nearly 800 million) worldwide by 2045. Sedentary behavior and increased adiposity are major risk factors for T2D. Cardiovascular disease is the leading cause of death in those with T2D, while diabetic microvascular disease, causing kidney disease, neuropathy, and retinopathy, contributes to T2D morbidity.

Physical activity is one of the most potent therapies in preventing/treating T2D and its complications. Mean daily steps is a proxy for physical activity, with even modest improvements in step count (i.e., +500 steps) associated with decreased T2D and mortality. However, adherence to regular physical activity remains low in T2D patients, with short-term decreases in daily step count associated with impaired glycemic control and T2D recurrence.

The investigators have developed an artificial intelligence (AI) language model (similar to ChatGPT), which can automatically generate coaching prompts to encourage physical activity by incorporating an individual's stage of change. The investigators will extend our research using the My Heart Counts (MHC) smartphone app to 1) validate the efficacy of the AI-generated prompts in patients with T2D and 2) perform a longer-term randomized crossover trial using the language model as a social accountability chatbot - encouraging participants to maintain their physical activity changes over months. The investigators hypothesize that my AI-assisted coaching prompts will significantly increase 1) mean daily step count by 500 steps in 1,000 adults recruited nationwide over a 7-day period, and 2) improve HbA1c and weight via long-term behavior change over a 24-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥18 years old, with a clinical diagnosis of T2D, able to read and understand English, and who are physically able to walk, will be included in our study

Exclusion Criteria:

* Criteria that fall outside of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Mean daily steps | 7 days and 24 weeks
  Mean daily steps over the course of an intervention week (aim 1) and 24 week period (aim 2).

SECONDARY OUTCOMES:
Change in weight | 24 Weeks
  Change in weight over the long term intervention (Aim 2)
Change in HbA1c | 24 Weeks
  Change in HbA1c over the long term intervention (Aim 2)
Weekly Active Minutes | 7 days and 24 Weeks
  Total weekly active minutes over the course of an intervention week (aim 1) and 24 week period (aim 2).

IPD SHARING:
Plan to Share IPD: No